CLINICAL TRIAL: NCT01478178
Title: Open-label, Single Arm, Safety and Tolerability Dose Escalation Study of VAL-083 in Patients With Recurrent Malignant Glioma
Brief Title: Safety Study of VAL-083 in Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kintara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLM-10-001
Record Dates: First submitted 2011-11-14; First posted 2011-11-23 (Estimated); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Glioma; Glioblastoma; Glioblastoma Multiforme; GBM; Brain Cancer
Keywords: Glioma; Glioblastoma; Glioblastoma multiforme; GBM; brain tumor; brain cancer; recurrent brain tumor; recurrent brain cancer; refractory brain tumor; refractory brain cancer; recurrent GBM; refractory GBM; recurrent glioma; refractory glioma; recurrent glioblastoma; refractory glioblastoma; recurrent glioblastoma multiforme; refractory glioblastoma multiforme; failed temodar; failed temozolomide; temodar refractory; temozolomide refractory; failed avastin; avastin refractory; failed bevacizumab; bevacizumab refractory; avastin failure; bevacizumab failure; temodar failure; temozolomide failure
MeSH Terms: conditions — Glioma; Glioblastoma; Brain Neoplasms | interventions — Dianhydrogalactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VAL-083 (Dianhydrogalactitol) (Experimental): VAL-083 given by intravenous infusion with a starting dose of 1.5 mg/m2 IV. Escalating doses to be administered in sequential dose cohorts.
  Interventions: Drug: VAL-083 (Dianhydrogalactitol)

INTERVENTIONS:
Drug: VAL-083 (Dianhydrogalactitol) — VAL-083 given by intravenous infusion with a starting dose of 1.5 mg/m2 IV. Escalating doses to be administered in sequential dose cohorts.

SUMMARY:
The purpose of this Phase 1/2, open-label, single-arm study is to determine the safety and the maximal tolerated dose (MTD) of VAL-083 in patients with recurrent malignant glioma. Pharmacokinetic (PK) properties will be explored and tumor responses to treatment will be evaluated.

DETAILED DESCRIPTION:
Recurrent glial tumors of the brain continue to be one of the most challenging malignancies to treat. Median survival for patients with recurrent disease is approximately 6 months for glioblastoma multiforme. Bevacizumab is used for treatment of recurrent disease; however patients who fail bevacizumab do not have many treatment options.

Metastases to the brain are the most common intracranial tumors in adults and occur ten times more frequently than primary brain tumors. It is estimated that 8 - 10% of cancer patients may develop symptomatic metastatic tumors in the brain. Systemic therapy is rarely used for primary treatment of brain metastases because many tumors that metastasize to the brain are not chemosensitive or have been already heavily pretreated with potentially effective agents, and poor penetration through the blood brain barrier is an additional concern.

Dianhydrogalactitol (DAG) rapidly penetrates both the cerebrospinal fluid (CSF) and the blood-brain barrier and accumulates in brain tissue. Clinical study of DAG in patients with GBM or with progressive secondary brain tumors is warranted. Patients with secondary brain metastases were allowed to enroll into the current protocol in Cohorts 2 and 3; however, enrollment ceased with Amendment 5 and will not be continued beyond Cohort 3.

This study will utilize a standard 3 + 3 dose escalation design, until the MTD or the maximum specified dose has been reached. In Phase 2, additional patients with GBM will be treated at the MTD (or other selected optimum Phase 2 dose) to measure tumor responses to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be greater than or equal to 18 years old.
* Histologically confirmed initial diagnosis of primary WHO Grade IV malignant glioma (glioblastoma), now recurrent; or Cohorts 2 and 3 only: progressive secondary brain tumor, has failed standard brain radiotherapy, and has brain tumor progression after at least one line of systemic therapy. Patients with progressive secondary brain tumors will not be enrolled under this protocol following the completion of Cohort 3.
* If GBM, previously treated for GBM with surgery and/or radiation, if appropriate, and must have failed both bevacizumab (Avastin) and temozolomide (Temodar), unless either or both are contraindicated.
* If GBM, greater than or equal to 12 weeks from radiotherapy, or 4 weeks if a new lesion, relative to the pre-radiation MRI, develops that is outside the primary radiation field.
* Cohorts 2 & 3 only: Patients with secondary brain tumors must be greater than or equal to 4 weeks from radiotherapy. Patients with progressive secondary brain tumors will not be enrolled under this protocol following the completion of Cohort 3.
* At least 4 weeks from last chemotherapy or bevacizumab (Avastin) therapy (6 weeks for nitrosourea or mitomycin C), or for chemotherapy regimes given continuously or on a weekly basis with limited potential for delayed toxicity, at least 2 weeks from last dose.
* At least 21 days or 5 half-lives (whichever is shorter) since prior investigational anti-cancer drugs. A minimum of 10 days between termination of the investigational drug and administration of DAG is required
* Recovered from all treatment-related toxicities to Grade 1 or less.
* Must have a Karnofsky performance status of > 50 with a predicted life expectancy of at least 12 weeks.
* Must have known MGMT methylation and IDH1 mutation status to be screened for study entry.

Exclusion Criteria:

* Current history of neoplasm other than the entry diagnosis. Patients with previous cancers treated and cured with local therapy alone may be considered with approval of the Medical Monitor.
* Evidence of leptomeningeal spread of disease.
* Evidence of recent hemorrhage on baseline MRI of the brain.
* Concurrent severe, intercurrent illness.
* History of severe cardiac disease.
* Significant vascular disease.
* History of stroke or transient ischemic attack within 6 months prior to beginning treatment.
* Concomitant medications that are known inducers of CYP.
* Concomitant medications that are strong inhibitors of cytochrome P450 and CYP3A up to 14 days before Cycle 1 Day 1 (pimozide, diltiazem, erythromycin, clarithromycin, and quinidine, and amiodarone up to 90 days before)
* Known to be HIV positive or to have an AIDS-related illness.
* Pregnant or breast feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-10; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose (MTD) | Study Day 35
  The determination of MTD will be based on analysis of tolerance data from the first cycle of therapy in each dose group.

SECONDARY OUTCOMES:
Evaluate tumor response in patients with recurrent malignant glioma | Every 60 days
  Tumor assessment every other treatment cycle, as long as patient continues to demonstrate response or stable disease and tolerates therapy.
Characterization of Cycle 1 plasma pharmacokinetics | Cycle 1: 0, 0.25, 0.5, 1, 2, 4, 6 hrs and immediately prior to Cycle 1, Day 2 dosing
  Plasma will be analyzed to estimate appropriate PK parameters (Cmax, Tmax, AUC, elimination half-life, drug clearance, mean residence time, and volume of distribution).

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Burris, M.D., Principal Investigator — Sarah Cannon Research Institute; Nashville, Tennessee 37203, USA; Manish Patel, M.D., Principal Investigator — Florida Cancer Specialists, Sarasota, Florida 34232, USA; Nicholas Butowski, M.D., Principal Investigator — University of California, San Francisco, 94143, USA; Sani Kizilbash, M.D., Principal Investigator — Mayo Clinic, Rochester, Minnesota 55905, USA; Gerald Falchook, M.D., Principal Investigator — Sarah Cannon Research Institute; Denver, Colorado 80218 USA
Locations (5):
- United States (5):
  - University of California, San Francisco, Division of Neuro-Oncology, San Francisco, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
The Clinical Study Report for this trial will be prepared and provided to U.S. F.D.A. as required by applicable regulatory requirement(s). Each participating trial investigator has been provided a copy their patient data captured in the electronic data base for this trial.